CLINICAL TRIAL: NCT05583734
Title: A Prospective Study of Conventional Bone Marrow Biopsies and Bone Marrow Biopsies Performed Through the Portomar(TM), Using a Modified PROMIS Pain Intensity Scale for Pain Assessment
Brief Title: A Prospective Study of Conventional Bone Marrow Biopsy Versus Portomar(TM) Biopsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aperture Medical Technology, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Study Number: 1339403
Record Dates: First submitted 2022-09-29; First posted 2022-10-18 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Self-controlled, prospective trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Portomar(TM) Device (Experimental): Portomar(TM) Device for bone marrow biopsy
  Subjects are self-controlled with one side having conventional biopsy and the other having the Portomar(TM) biopsy.
  Interventions: Device: Portomar(TM) Device

INTERVENTIONS:
Device: Portomar(TM) Device — Portomar(TM) access device for bone marrow biopsy

SUMMARY:
This is a self-controlled, prospective trial. The objective of this trial is to evaluate the efficacy and safety of the Portomar(TM) device for bone marrow biopsy.

DETAILED DESCRIPTION:
This is a self-controlled, prospective trial. Subjects will undergo conventional bone marrow biopsy compared to bone marrow biopsy with the Portomar(TM) device. Subjects will be evaluated at multiple time points comparing the two biopsies. Data through the 6 month time point will be used for Regulatory Submission to the FDA. Additionally subjects will be followed for two years post enrollment.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with a previous bone marrow disorder diagnosis who will require multiple bone marrow biopsies over the course of their treatment, for example patients with plasma cell dyscrasia or leukemia.

  * Men and non-pregnant women of age ≥ 21 years with ECOG performance status ≤ 2.
  * Any hematologic (platelets above 50, ANC > 1.0, hemoglobin > 7), renal (patients not on dialysis), or hepatic (patients with bilirubin below 2.5) function status suitable to undergo port implantation and subsequent bone marrow biopsies.
  * Patients must be able to understand and be willing to sign a voluntary informed consent form and agree to compliance with the protocol schedule; with the knowledge that they may withdraw consent at any time without impact on future medical care.

Exclusion Criteria:

* • Patients with any other ongoing, concomitant, comorbid illness including but not limited to uncontrolled diabetes, NYHA class III or worse heart failure, uncontrolled coronary artery disease/arrhythmia.

  * Patients unable to comply with the study schema.
  * Confirmed pregnancy at time of screening or on implantation day prior to anesthesia/sedation.
  * Patients unable to come off of anticoagulation medications for their procedure.
  * Patients with active infection.
  * Patients with < 0.5 cm or > 2.5 cm of soft tissue between screw head and skin at the target site of implantation. This is based on the patient's prior imaging studies (i.e. CT/MR or ultrasound imaging).
  * Patient has contra-indication to conscious sedation or anesthesia services
  * Patients who have had prior bone marrow biopsy within 2 weeks of the study biopsy.
  * Patients with coagulopathy such that INR cannot be corrected < 2.0.
  * Patients who are prisoners or wards of the court.
  * Patients with alcohol or substance abuse disorder defined by DSM V criteria.
  * Patients with the diagnosis of a major psychiatric disorder such as schizophrenia or major depression defined by the DSM-V criteria.
  * Patients with osteoporosis defined as L1 vertebrae bone density lower than 90 Hounsfield units

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Day of bone marrow biopsy (approximately 1 month after Portomar(TM) placement)
  Pain Comparison- The scale used to assess pain is a modified National Cancer Institute (NCI) Patient Reported Outcome Measurement Information System (PROMIS). Patients are asked to rate their pain intensity from 0 (no pain)-10 (worst pain ever) comparing the bone marrow biopsy performed with the Portomar(TM) device and a standard bone marrow biopsy. The endpoint will be the proportion of patients experiencing at least a 2 point improvement in score between Portomar(TM) and standard biopsy.
Portomar(TM) pain intensity | Day of placement (beginning of study)
  Pain related to Portomar(TM) will be assessed using the same modified NCI PROMIS Scale. The endpoint is the proportion of patients experiencing severe pain (>8).
Portomar(TM) pain intensity | 1 day after study begins with Portomar(TM) placement
  Pain related to Portomar(TM) will be assessed using the same modified NCI PROMIS
Portomar(TM) pain intensity | 2 days after study begins with Portomar(TM) placement
  Pain related to Portomar(TM) will be assessed using the same modified NCI PROMIS
Portomar(TM) pain intensity | 7 days after study begins with Portomar(TM) placement
  Pain related to Portomar(TM) will be assessed using the same modified NCI PROMIS
Portomar(TM) pain intensity | 14 days after study begins with Portomar(TM) placement
  Pain related to Portomar(TM) will be assessed using the same modified NCI PROMIS
Portomar(TM) pain intensity | 30 days after study begins with Portomar(TM) placement
  Pain related to Portomar(TM) will be assessed using the same modified NCI PROMIS
Portomar(TM) pain intensity | 90 days after study begins with Portomar(TM) placement
  Pain related to Portomar(TM) will be assessed using the same modified NCI PROMIS

SECONDARY OUTCOMES:
Safety Events | Study duration, approximately 2 years
  Adverse events
Satisfaction Score | Day of placement and every time a bone marrow biopsy is performed using the Portomar(TM) device for study duration approximately 2 years
  Patient and practitioner satisfaction questionnaires
Pain Score | Study duration (approximately 2 years) at all bone marrow biopsies with Portomar(TM)
  Pain from Portomar(TM) and bone marrow biopsies. The modified PROMIS scale 0-10 will be used.
Specimen-Core Biopsy | Study duration (approximately 2 years) at all bone marrow biopsied performed with Portomar(TM)
  Adequacy. This will be judged by the proportion of biopsies at least 1.2 cm length.
Specimen-Aspirate | Study duration (approximately 2 years) at all bone marrow biopsied performed with Portomar(TM)
  Adequacy This will be judged by the proportion of aspirations with at least 1 spicule seen.
Time | Study duration (approximately 2 years) at all bone marrow biopsied performed with Portomar(TM)
  Time from needle anesthetic to sample acquired. Comparison of conventional vs. Portomar(TM).

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Sheth, Principal Investigator — MD Anderson
Locations (1):
- MD Anderson, Houston, Texas, United States